CLINICAL TRIAL: NCT00890552
Title: A Pilot Study of Lenalidomide, Melphalan and Dexamethasone in AL Amyloidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Stanley L Schrier, Professor of Medicine, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15213; RV-AMYL-PI-0375 (Other: Celgene Reference number); SU-09192008-1300 (Other: Stanford University); HEM0010 (Other: OnCore)
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Results first posted 2017-03-22 (Actual); Last update posted 2017-03-22 (Actual); Status verified 2017-02

CONDITIONS: Leukemia; Amyloidosis
MeSH Terms: conditions — Leukemia; Amyloidosis | interventions — Lenalidomide; Melphalan; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide+Melphalan+Dexamethasone (Experimental): Patients received lenalidomide 10 mg/day orally on days 1-21, melphalan 0.18 mg/kg orally on days 1-4, and dexamethasone 40 mg orally once weekly of a 28-day cycle (MDR treatment).
  Interventions: Drug: Lenalidomide; Drug: Melphalan; Drug: Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide is a a derivative of thalidomide.
  Orally-administered lenalidomide 10 mg will be taken daily on days 1 to 21 of 28-day cycle.
  Other Names: Revlimid; L04AX04
Drug: Melphalan — Melphalan is a phenylalanine derivative of mechlorethamine.
  Orally-administered melphalan 0.18 mg/kg will be taken on days 1 to 4 of a 28-day cycle
  Other Names: Alkeran; Evomela; Sarcolysin; L-phenylalanine mustard (L-PAM); 4-[Bis(2-chloroethyl)amino]-L-phenylalanine
Drug: Dexamethasone — Dexamethasone is an anti-inflammatory and immunosuppressant steroid medication.
  Orally-administered dexamethasone 40 mg orally once weekly of a 28-day cycle
  Other Names: Intensol; Decadron; Baycadron; Dexpak® Taperpak; Maxidex (dexamethasone ophthalmic suspension); Ozurdex (dexamethasone intravitreal implant)

SUMMARY:
This open-label trial will evaluate the use of lenalidomide; melphalan; and dexamethasone (MDR) to treat newly diagnosed or relapsed AL amyloidosis, over the course of nine 28-day cycles.

DETAILED DESCRIPTION:
The study will evaluate the 3-drug combination of lenalidomide; melphalan; and dexamethasone (MDR) as the absence of disease progression or toxicity, patients will complete nine 28-day cycles of MDR therapy, with the option of continuing treatment with lenalidomide as single-agent. Patients received up to nine cycles of treatment, with the option to continue on lenalidomide as a single agent if they responded to treatment.

ELIGIBILITY:
INCLUSION CRITERIA

* Newly diagnosed or relapsed AL amyloidosis
* Biopsy-proven amyloidosis with evidence of an underlying plasma cell dyscrasia

  * abnormal clonal dominance of plasma cells in the bone marrow
  * detection of a monoclonal gammopathy by immunofixation electrophoresis of serum and/or urine
  * an abnormal serum free light chain or ratio, or AL fibrils seen on biopsy)
* Measurable disease defined by an abnormal serum-free light chain or monoclonal protein by immunofixation

  * proteinuria ≥ 0.5 g/day, cardiac involvement with interventricular septal thickness ≥ 15 mm
  * hepatomegaly in the absence of congestive heart failure with elevated alkaline phosphatase
* Age ≥ 18 years at the time of signing the informed consent form.
* All previous cancer therapy must have been discontinued at least 4 weeks prior to treatment in this study
* ECOG performance status of ≤ 3 at study entry
* Laboratory test results:

  * Absolute neutrophil count ≥ 1.0 x 10e9 / L
  * Platelet count ≥ 75 x 10e9 / L
  * Creatinine clearance ≥ 15 mL/ minute
  * Total bilirubin ≤ 2-fold upper limits of normal
* Disease-free of prior malignancies (excluding multiple myeloma) for ≥ 3 years with exception of:

  * currently treated basal cell
  * squamous cell carcinoma of the skin
  * carcinoma "in situ" of the cervix or breast.
* Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test
* Females of childbearing potential must either:

  * commit to continued abstinence from heterosexual intercourse
  * acceptable methods of birth control and agree to ongoing pregnancy testing
* Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy
* All study participants must be registered into the mandatory RevAssist program, and able to comply with its requirements
* Able to take aspirin (81 mg) daily • Understand and voluntarily sign an informed consent form
* Able to adhere to the study visit schedule and other protocol requirements

EXCLUSION CRITERIA

* Any serious medical condition that would prevent the subject from signing the informed consent form
* Pregnant
* breast-feeding females
* Use of any other experimental drug or therapy within 28 days of baseline
* Known hypersensitivity to thalidomide
* Erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs
* Any prior use of lenalidomide
* Concurrent use of other anti-cancer agents or treatments
* Known positivity for human immunodeficiency virus HIV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2009-04; Primary Completion 2012-08 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L Schrier, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University Cancer Institute, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palladini G, Dispenzieri A, Gertz MA, Kumar S, Wechalekar A, Hawkins PN, Schonland S, Hegenbart U, Comenzo R, Kastritis E, Dimopoulos MA, Jaccard A, Klersy C, Merlini G. New criteria for response to treatment in immunoglobulin light chain amyloidosis based on free light chain measurement and cardiac biomarkers: impact on survival outcomes. J Clin Oncol. 2012 Dec 20;30(36):4541-9. doi: 10.1200/JCO.2011.37.7614. Epub 2012 Oct 22. PMID 23091105
- [Result] Dinner S, Witteles W, Afghahi A, Witteles R, Arai S, Lafayette R, Schrier SL, Liedtke M. Lenalidomide, melphalan and dexamethasone in a population of patients with immunoglobulin light chain amyloidosis with high rates of advanced cardiac involvement. Haematologica. 2013 Oct;98(10):1593-9. doi: 10.3324/haematol.2013.084574. Epub 2013 May 28. PMID 23716538

RESULTS

PARTICIPANT FLOW:
Groups:
- Lenalidomide, Melphalan and Dexamethasone (MDR): The 3-drug combination of orally-administered lenalidomide; melphalan; and dexamethasone (MDR) will be administered as nine 28-day cycles, with the option of continuing treatment with lenalidomide as single-agent.
  Lenalidomide: Orally-administered lenalidomide 10 mg will be taken daily on days 1 to 21 of 28-day cycle. Lenalidomide is a a derivative of thalidomide.
  Melphalan: Orally-administered melphalan 0.18 mg/kg will be taken on days 1 to 4 of a 28-day cycle. Melphalan is a phenylalanine derivative of mechlorethamine.
  Dexamethasone: Orally-administered dexamethasone 40 mg will be taken on days 1; 8; 15; and 22 of a 28-day cycle. Dexamethasone is an anti-inflammatory and immunosuppressant steroid medication.
Period: Enrollment and Pre-treatment
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Started | 25
Completed | 24
Not Completed | 1
Not completed — Death/ lost to follow up | 1
Period: On-treatment
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Started | 24
Completed | 14
Not Completed | 10
Not completed — Early prog disease/ death | 10

BASELINE CHARACTERISTICS:
Population: Lenalidomide-naïve adults with biopsy-proven amyloidosis manifested as measurable disease, ECOG ≤ 3
Groups:
- Lenalidomide, Melphalan and Dexamethasone (MDR): The 3-drug combination of orally-administered lenalidomide; melphalan; and dexamethasone (MDR) will be administered as nine 28-day cycles, with the option of continuing treatment with lenalidomide as single-agent.
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 67 [52 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 1
ECOG Performance Status (PS) [Number; unit: participants] — ECOG Performance Status. PS 0 = Fully active, able to carry on all pre-disease performance without restriction.
  PS 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  PS 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours. PS 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours..
  participants
    ECOG PS 1 | 12
    ECOG PS 2 | 9
    ECOG PS 3 | 4
Hematologic disease burden [Number; unit: Percentage of participants]
  Kappa free light chain (%) | 20
  Lambda free light chain (%) | 80

OUTCOME MEASURES:

1. Primary Outcome: Hematologic Response Rate
Description: At the end of each treatment cycle (4 weeks), hematologic response rate as assessed. Hematologic response was considered to be amyloid complete response (normal FLC ratio and negative serum and urine immunofixation); very good partial response (difference between involved and uninvolved FLCs [dFLC] < 40 mg/L); or partial response (dFLC decrease > 50%).
Time Frame: 8 weeks
Population: Subjects completing at least one full cycle of study treatment
Measure: Number; unit: participants
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Number analyzed (Participants) | 24
participants
  Complete Response (CR) | 2
  Very good Partial Response (VGPR) | 4
  Partial Response (PR) | 8
  No Response (NR) | 9
  Response not evaluable | 1

2. Secondary Outcome: Overall Survival (OS)
Description: Participants alive 12 months after starting MDR treatment.
Time Frame: 12 months
Population: All subjects receiving MDR treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Number analyzed (Participants) | 24
percentage of participants | 58

3. Secondary Outcome: Event-free Survival (EFS)
Description: Assessed as the median value for EFS 12 months after starting MDR treatment
Time Frame: 12 months
Population: All participants starting MDR treatment
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Number analyzed (Participants) | 14
months | 3.15 [0.25 to 12]

4. Secondary Outcome: Duration of Response
Description: Assessed as the median value for the time from first partial response until progression; death; or last follow-up.
Time Frame: 32 months
Population: All participants who achieved at least a partial response (9 subjects were not included due to not having any response)
Measure: Median (Full Range); unit: months
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Number analyzed (Participants) | 14
months | 9.1 [0 to 31.25]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Lenalidomide, Melphalan and Dexamethasone (MDR)
Serious Adverse Events (participants affected / at risk) | 19/25
Other Adverse Events (participants affected / at risk) | 23/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Melphalan and Dexamethasone (MDR) (N=25)
Hyponatremia (Metabolism and nutrition disorders) | 3
Atrial fibrillation (Cardiac disorders) | 4
Febrile neutropenia (Infections and infestations) | 1
Hemorrhage (Gastrointestinal disorders) | 2
Death (General disorders) | 7
Dehydration (Gastrointestinal disorders) | 2
Syncope (General disorders) | 4
Anemia in Neoplastic disease (Blood and lymphatic system disorders) | 1
Primary Amyloidosis (Metabolism and nutrition disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Altered mental status (Psychiatric disorders) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Edema (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 1
Hypoglycemia (Blood and lymphatic system disorders) | 1
Hypovolemia (Blood and lymphatic system disorders) | 1
Renal failure (Metabolism and nutrition disorders) | 1
Pneumonia (Infections and infestations) | 1
Atrial flutter (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide, Melphalan and Dexamethasone (MDR) (N=25)
Anorexia (Gastrointestinal disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Bone and Blood Marrow (Blood and lymphatic system disorders) | 5
Hypocalcemia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Creatinine (Metabolism and nutrition disorders) | 3
Dermatology (Skin and subcutaneous tissue disorders) | 2
Diarrhea (Gastrointestinal disorders) | 5
Distension/bloating (Gastrointestinal disorders) | 3
Dizziness (Nervous system disorders) | 7
Dry mouth (Gastrointestinal disorders) | 3
Dysphagia (Respiratory, thoracic and mediastinal disorders) | 10
Edema: limbs (Infections and infestations) | 11
Fatigue (General disorders) | 16
Fever (General disorders) | 5
Gastrointestinal (Gastrointestinal disorders) | 8
Hyperglycemia (Metabolism and nutrition disorders) | 3
Hematoma (Hepatobiliary disorders) | 2
Hemoglobin (Hepatobiliary disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 6
Hypotension (Cardiac disorders) | 3
Infection (Infections and infestations) | 11
INR (Blood and lymphatic system disorders) | 2
Insomnia (General disorders) | 4
Leukocytes (Blood and lymphatic system disorders) | 2
Mood alteration- Anxiety (General disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 6
Neutrophils/granulocytes (Blood and lymphatic system disorders) | 4
Pain (General disorders) | 12
Platelets (Blood and lymphatic system disorders) | 18
Hypokalemia (Metabolism and nutrition disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 11
Hyponatremia (Metabolism and nutrition disorders) | 5
Thrombotic microangiopathy (Cardiac disorders) | 2
Vision-blurred (Eye disorders) | 2
Vomitting (Gastrointestinal disorders) | 2
weight loss (Gastrointestinal disorders) | 5
Alkaline phosphatase (Metabolism and nutrition disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
AST, SGOT (Metabolism and nutrition disorders) | 1
Auditory/Ear (Ear and labyrinth disorders) | 1
Hyperbilirubinemia (Metabolism and nutrition disorders) | 1
Coagulation (Blood and lymphatic system disorders) | 1
Cystitis (Renal and urinary disorders) | 1
Dehydration (General disorders) | 1
abscess (Infections and infestations) | 1
Dry eye syndrome (Eye disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Edema: head and neck (Blood and lymphatic system disorders) | 1
Edema: trunk/genital (Blood and lymphatic system disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Hearing loss (Ear and labyrinth disorders) | 1
Lymphatics (Blood and lymphatic system disorders) | 1
Depression (Psychiatric disorders) | 1
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Neuropathy: motor (Nervous system disorders) | 1
Ocular/Visual (Eye disorders) | 1
Petechiae/purpura (Skin and subcutaneous tissue disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Rigors/chills (General disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Sweating (Skin and subcutaneous tissue disorders) | 1
dysarthria (General disorders) | 1
Wound complication (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes